CLINICAL TRIAL: NCT01851798
Title: Postoperative Home Sleep Test Changes in Ambulatory Surgical Patients With and Without Obstructive Sleep Apnea: A Prospective Clinical Trial
Brief Title: Evaluation of Sleep Disordered Breathing Following Ambulatory Surgery
Status: Terminated | Type: Observational
Why Stopped: Staffing changes precluded sleep study interpretation
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, Arlene Hudson, Assistant Professor of Anesthesiology, Walter Reed National Military Medical Center
Other Study IDs: WRNMMC IRB#384867
Record Dates: First submitted 2013-05-08; First posted 2013-05-10 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Sleep Disordered Breathing
Keywords: OSA; Sleep disordered breathing; anesthesia; ambulatory orthopedic surgery
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ambulatory orthopedic surgery patients with OSA: ambulatory orthopedic surgery patients with home sleep test preoperative AHI => 5
  Interventions: Other: Home sleep test administered to all enrolled subjects
- ambulatory orthopedic surgery patients without OSA: ambulatory orthopedic surgery patients with home sleep test preoperative AHI < 5
  Interventions: Other: Home sleep test administered to all enrolled subjects

INTERVENTIONS:
Other: Home sleep test administered to all enrolled subjects

SUMMARY:
Obstructive sleep apnea (OSA) is a relatively common medical condition that includes upper-airway obstruction and consequent cessation of breathing during sleep with significant associated other medical problems. The time period around surgery has been demonstrated to be an independent risk factor for various complications but the mechanism is not well understood.

This protocol proposes to study the fundamental question of what changes occur in the postoperative setting to ambulatory patients with and without OSA by administering a validated "STOP-BANG" screening questionnaire and conducting preoperative and postoperative Home Sleep Testing (HST). In doing so, critical evidence shall be gained in the understanding of postoperative sleep disorder breathing changes associated with surgery and anesthesia. With evidence, sound perioperative management recommendations and policy may be developed to assist with caring for this large and at risk surgical population.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a highly prevalent syndrome of upper-airway obstruction and consequent cessation of respiration during sleep. Associated complications include impairment in the cardiovascular and cerebrovascular, neurological and endocrine systems. There is growing concern that the perioperative period may acutely worsen existing OSA or potentially induce sleep disordered breathing in susceptible individuals. Indeed, the presence of OSA has been shown to be an independent risk factor for perioperative complications. The mechanism for this perioperative risk, however, has yet to be fully elucidated.

This study proposes to investigate the relationship between surgical anesthesia and OSA with an observational prospective single-blinded investigation. A sample of 600 adult female and male orthopedic surgery patients scheduled for elective ambulatory orthopedic surgery at WRNMMC will be enrolled. Study subjects shall undergo an unattended Home Sleep Test (HST) the night before surgery followed by surgery and anesthesia as determined by the surgical team unchanged by study participation. Following the surgical procedure and anesthesia, the study subject will undergo a series of two additional HSTs on the first night following surgery and again on post-operative night three and complete a postoperative questionnaire including a validated screening questionnaire and information pertaining to postoperative pain and medication use.

Qualitative and quantitative analysis will be performed on the data. The prevalence in the ambulatory orthopedic population of screening positive with the STOP-BANG questionnaire, a validated Obstructive Sleep Apnea (OSA) screening tool, will be determined as well as the prevalence of OSA diagnosed by the preoperative Home Sleep Test (HST). The analysis of the HST data will be blinded as to OSA status, if known, and screening results using the validated "STOP-BANG" screening questionnaire. There are several additional research questions posed in this observational prospective single-blinded clinical study to determine if OSA, as defined by apnea-hypopnea index (AHI), is a significant factor in adverse events associated with ambulatory orthopedic surgery. First, a study sample size of 600 was selected to provide 82% power to detect a significant difference in unplanned admissions between patients with OSA (estimated at 20% of the surgical orthopedic population) and without OSA. This assumes 10% of patients without OSA experience unplanned admissions compared with 20% of patients with OSA. Other adverse perioperative events to be examined include difficult intubations, upper airway obstruction after extubation, bronchospasm, laryngospasm, arrhythmia such as atrial fibrillation, and need for mechanical ventilation

Additional questions to be examined include if surgery and anesthesia, the specific anesthetic technique, intraoperative sedative use, or postoperative sedative use is associated with any Home Sleep Test (HST) parameter (AHI, Oxygen Desaturation Index (ODI), pulse oximetry (SpO2) nadir, or percentage of time SpO2<90%). Paired t-tests will be used to perform the analyses except for the question of anesthetic technique for which analysis of variance followed by Tukey's post-hoc multiple comparisons will be employed.

Lastly is the clinically relevant question addressing whether there is a difference between patients who screen as high risk for OSA and those who screen as low risk for OSA with regard to pre and postoperative AHI, ODI, SpO2 nadir, or percentage of time SpO2<90%? High- and low-risk patients per the screening instrument will be compared using t-tests for independent samples.

Ultimately understanding the relationship between surgical anesthesia and OSA may be used to risk stratify patients, identify those at an increased risk for perioperative complications, or potentially aid in determining perioperative management plans.

ELIGIBILITY:
Inclusion Criteria:

* Male and female military health care beneficiaries between the ages of 18 and 85 years presenting for elective ambulatory orthopedic surgery at WRNMMC main operating room.
* American Society of Anesthesiologist physical classification (ASA) I-II
* Scheduled for elective ambulatory orthopedic surgery
* Patients English speaking and capable of providing informed consent.

Exclusion Criteria:

* Patients who are pregnant or breast-feeding at the time of the procedure. Pregnancy will be ruled out by day of surgery urine human chorionic gonadotropin (HCG) when appropriate.
* Chronic opioid, benzodiazepine, pregabalin, or other sedating medication users
* Chronic alcohol users (defined by daily or greater use upon standard anesthesia preoperative interview)
* Patients who require home oxygen use
* Patients who have a tracheostomy
* Patients who decline to participate.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ambulatory orthopedic surgery patients presenting to Walter Reed National Military Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Unplanned hospital admission | First three post operative days

SECONDARY OUTCOMES:
Prevalence of OSA in orthopedic ambulatory surgical population | Determined by home sleep test on night before surgery over study duration expected to be 2-3 years
  Prevalence of OSA in study population will be evaluated by preoperative home sleep test. The number of enrolled subject who have a home sleep test Apnea Hypopnea Index (AHI)=>5 will be considered positive. Prevalence will be determined by the percent of subjects who test positive of all those enrolled over the study period.

OTHER OUTCOMES:
Significant Change in Apnea-Hypopnea Index | Night before surgery to the second post operative night

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Hudson, MD, Principal Investigator — Walter Reed National Military Medical Center and Uniformed Services University of the Health Sciences
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Hudson AJ, Walter RJ, Flynn J, Szpisjak DF, Olsen C, Rodgers M, Capaldi VF 2nd, McDuffie B, Lettieri CJ. Ambulatory Surgery Has Minimal Impact on Sleep Parameters: A Prospective Observational Trial. J Clin Sleep Med. 2018 Apr 15;14(4):593-602. doi: 10.5664/jcsm.7052. PMID 29609705